CLINICAL TRIAL: NCT00046111
Title: A Study to Determine the Bioequivalence of an Oral Formulation of Topotecan Containing the Drug Substance Manufactured by New Process Relative to the Current Study Formulation of Topotecan in Patients With Advanced Solid Tumors
Brief Title: A Bioequivalence Study of Two Oral Formulations of Topotecan in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 104864-A/565
Record Dates: First submitted 2002-09-19; First posted 2002-09-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer, Small Cell; Solid Tumor Cancer
Keywords: oral; Bioequivalence; Hycamtin; Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

ARMS (1):
- Primary Group (Experimental): 40 subjects on medium doses of Topotecan and tested for bioequivalence for 4 weeks.
  Interventions: Drug: topotecan

INTERVENTIONS:
Drug: topotecan — A topoisomerase I inhibitor used for ovarian and lung cancer treatment

SUMMARY:
The purpose of this study is to compare two capsules of topotecan made by slightly different methods. This will be done by giving the drug made by the two different methods to patients orally and testing blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with confirmed advanced solid tumors.
* No prior chemotherapy within 5 years of the diagnosis of SCLC (small cell lung cancer).
* At least 4 weeks since last chemotherapy, radiotherapy, biologic therapy or surgery.
* Laboratory criteria: Patients must have adequate bone marrow reserve and adequate kidney and liver function.

Exclusion criteria:

* Women who are pregnant or lactating.
* Patients of child bearing potential refusing to practice adequate contraception.
* Patients with uncontrolled vomiting.
* Active infection.
* Patients with clinical evidence of any gastrointestinal (GI) conditions which would alter GI absorption or GI motility.
* Patients requiring treatment with cyclosporin A.
* Severe medical problems other than the cancer, that would limit the ability of the patient to follow study guidelines or expose the patient to extreme risk.
* Ongoing or planned chemotherapy, immunotherapy, radiotherapy, or investigational therapy for cancer treatment.
* Use of investigational drug within 30 days prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2001-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To determine the bioequivalence of new formulation (test) of oral topotecan relative to the current Phase III formulation (reference) of oral topotecan by comparing AUC in patients with advanced solid tumors. | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (4):
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Ottawa, Ontario, Canada